CLINICAL TRIAL: NCT05471726
Title: Improving Post-discharge Antimicrobial Use: a Multicenter Stepped Wedge Trial Study
Brief Title: Improving Post-discharge Antimicrobial Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB 202109288
Record Dates: First submitted 2022-07-13; First posted 2022-07-25 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Infections
Keywords: antibiotic prescriptions; hospital discharge; antibiotic stewardship
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Stepped-wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective audit-and-feedback at discharge (Experimental): When hospitals are in the intervention arm, they will perform the audit-and-feedback process focused on patients receiving antimicrobials who have an anticipated discharge.
  Interventions: Behavioral: Prospective audit-and-feedback
- Standard of care (No Intervention): When hospitals are in the control arm, they will not perform a stewardship process that focuses on hospital discharge.

INTERVENTIONS:
Behavioral: Prospective audit-and-feedback — The stewardship team will review patients who are on antibiotics, have an uncomplicated infection, and are eligible to continue antibiotics after discharge. Any recommendations from the stewardship team about optimizing antibiotic therapy will be presented to the primary prescriber in real-time with the goal of improving antibiotic selection and duration at hospital discharge.
  Arms: Prospective audit-and-feedback at discharge

SUMMARY:
One in five hospitalized patients is prescribed an antimicrobial at the time of discharge, and a large proportion of these post-discharge antimicrobials are unnecessary. The investigators will evaluate a novel method for reviewing post-discharge antimicrobial prescriptions in real-time with the goal of improving antimicrobial selection and duration.

DETAILED DESCRIPTION:
Antimicrobial stewardship programs (ASPs) work to improve antibiotic prescribing within hospitals. ASPs often restrict their activities to inpatient antimicrobial-prescribing. However, at least 40% of all antimicrobial exposure associated with an acute-care hospital stay is prescribed at the time of hospital discharge (i.e., post-discharge). Post-discharge antimicrobials mediate clinical outcomes after discharge and may facilitate the spread of antimicrobial resistance.

Several studies have shown that post-discharge antimicrobial use is often inappropriate. For example, using national VA data, the investigators found that 61% of fluoroquinolone treatment days were prescribed at hospital discharge; manual chart reviews at 9 hospitals found that 40% of these post-discharge fluoroquinolone prescriptions were either unnecessary or sub-optimal. Other studies have found that 53-79% of all post-discharge antimicrobials are either unnecessary or sub-optimal.

Post-discharge antimicrobials are an important target for antimicrobial stewardship. However, inpatient stewardship metrics do not capture post-discharge antimicrobials and ASPs frequently do not evaluate these prescriptions. A 2016 VA survey found that less than 50% of hospitals routinely reviewed targeted antimicrobials at discharge. According to a 2016 survey in Michigan, only 17% of 48 hospitals had a process for reviewing outpatient antimicrobial orders at discharge.

It is unclear how inpatient stewardship resources can be effectively leveraged to improve post-discharge antimicrobial use. If the goal is to improve post-discharge antimicrobial use, a potentially effective strategy may be an audit-and-feedback process focused solely on prescriptions for patients who will soon be discharged. In this trial, the investigators will evaluate the feasibility and effectiveness of such a process.

ELIGIBILITY:
Inclusion Criteria:

--The local stewardship team agrees to implement the discharge stewardship intervention on at least one inpatient service or ward.

Exclusion Criteria:

--The hospital already has an audit-and-feedback process in place that focuses on antimicrobial prescribing at hospital discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All patients on a participating inpatient service at the participating hospitals will be included, regardless of gender, race, or age.
Enrollment: 10 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Post-discharge antibiotic length of therapy | Every 2-week-period through study completion (48 weeks total)
  The primary outcome will be post-discharge antimicrobial length of therapy (LOT) per 100 admissions. The investigators will calculate this by adding post-discharge LOT across all patients on the participating services and dividing by the number of patient-admissions discharged from those services during the study period.

SECONDARY OUTCOMES:
Inpatient antibiotic length of therapy | Every two-week period through study completion (48 weeks total)
  Inpatient antibiotic LOT will be calculated by adding inpatient LOT across all patients on the participating services and dividing by the number of patient-admissions discharged from those services during the study period.
Percentage of participants with hospital readmission | 30 days from discharge
  Hospital readmissions reflect the need for (re) admission to an acute-care bed at a participating facility for any indication within 30 days of the patient's discharge.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Richard Roudebush VA Medical Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Barnes Jewish Hospital and affiliated hospitals, St Louis, Missouri
  - Audie L Murphy VA Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
All data will be aggregated to the hospital-level without including patient identifiers. This is a requirement for transmitting data across the institutions participating in this trial.

REFERENCES:
- [Derived] Livorsi DJ, Thompson AM, Green MS, Hoelscher AC, Chu KK, Neuner E, Burnett Y, Hopkins T, Walter E, Dave R, Tripathi R, Lohmar H, Dysangco A, Percival K, Ince D, Kolkmeyer J, Newland H, Hendrix MJ, Clore G, Poe C, O'Shea A, Tholany J, Prasidthrathsint K, Rachmiel E, Bongu J, Bewley A, Hsueh K. Prospective Audit and Feedback by Antibiotic Stewardship Teams to Reduce Antibiotic Overuse at Hospital Discharge: A Stepped-Wedge Cluster-Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2549655. doi: 10.1001/jamanetworkopen.2025.49655. PMID 41511774

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT05471726/Prot_SAP_000.pdf